CLINICAL TRIAL: NCT01209260
Title: Transseptal Needle Versus Radiofrequency Energy for Left Atrial Access (TRAVERSE-LA): A Randomized Controlled Trial
Brief Title: Transseptal Needle Versus Radiofrequency Energy for Left Atrial Access
Acronym: TRAVERSE-LA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Baylis Medical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MarcusHsu
Record Dates: First submitted 2010-09-09; First posted 2010-09-27 (Estimated); Results first posted 2014-01-28 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-01

CONDITIONS: Heart Diseases
Keywords: Transseptal Puncture; Radiofrequency Energy; Left Atrium Access; Left Atrial Catheterization; Ablation; Transseptal Catheterization; Electrocautery; Catheter Ablation; Atrial Fibrillation
MeSH Terms: conditions — Heart Diseases; Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiofrequency energy needle (Experimental): Radiofrequency energy needle for transseptal access
  Interventions: Device: Radiofrequency energy needle
- Mechanical needle (Active Comparator): Mechanical (Brockenbrough) needle for transseptal access
  Interventions: Device: Mechanical Needle

INTERVENTIONS:
Device: Radiofrequency energy needle — Radiofrequency energy needle for transseptal access
  Other Names: Baylis Medical Inc. transseptal needle; NRG RF transseptal needle
  Arms: Radiofrequency energy needle
Device: Mechanical Needle — Mechanical needle for transseptal access
  Other Names: Brockenbrough Needle
  Arms: Mechanical needle

SUMMARY:
This is a randomized controlled trial examining whether a mechanical needle versus a needle that uses radiofrequency energy is better at puncturing through a thin wall in the heart (called "transseptal puncture") as measured by procedure time, during an electrical procedure/study of the heart .

DETAILED DESCRIPTION:
Transseptal puncture is a commonly performed procedure allowing access to the left atrium for catheter ablation. Historically, a conventional Brockenbrough needle has been used for this procedure to mechanically puncture the fossa ovalis, which has been well described in the literature.1, 2 Although generally safe, serious complications such as perforation of the atrial wall or aorta can occur.3, 4

Previous studies have evaluated the feasibility and safety of radiofrequency (RF) energy applied to a conventional needle as a technique to access the left atrium, particularly in patients with a repeat procedure, fibrotic septum or aneurysmal septum.5, 6 As a result of this earlier work, a special proprietary device has been designed. The NRG RF needle (Baylis Medical Inc., Montreal, Canada), uses radiofrequency energy emitted from the needle tip to aid in transseptal access. Despite limited literature to support its superiority and safety7-9compared to the conventional approach, the new device has become adopted in some electrophysiology procedures involving a transseptal puncture.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing radiofrequency ablation within the left atrium through a transseptal approach
* Patients greater than 18 years of age

Exclusion Criteria:

* Patients unable to grant informed, written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Marcus, MD, Principal Investigator — University of California, San Francisco; Jonathan Hsu, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] ROSS J Jr, BRAUNWALD E, MORROW AG. Transseptal left atrial puncture; new technique for the measurement of left atrial pressure in man. Am J Cardiol. 1959 May;3(5):653-5. doi: 10.1016/0002-9149(59)90347-9. No abstract available. PMID 13649591
- [Background] B-Lundqvist C, Olsson SB, Varnauskas E. Transseptal left heart catheterization: a review of 278 studies. Clin Cardiol. 1986 Jan;9(1):21-6. doi: 10.1002/clc.4960090105. PMID 3943231
- [Background] Roelke M, Smith AJ, Palacios IF. The technique and safety of transseptal left heart catheterization: the Massachusetts General Hospital experience with 1,279 procedures. Cathet Cardiovasc Diagn. 1994 Aug;32(4):332-9. doi: 10.1002/ccd.1810320409. PMID 7987913
- [Background] De Ponti R, Cappato R, Curnis A, Della Bella P, Padeletti L, Raviele A, Santini M, Salerno-Uriarte JA. Trans-septal catheterization in the electrophysiology laboratory: data from a multicenter survey spanning 12 years. J Am Coll Cardiol. 2006 Mar 7;47(5):1037-42. doi: 10.1016/j.jacc.2005.10.046. Epub 2006 Feb 9. PMID 16516090
- [Background] Bidart C, Vaseghi M, Cesario DA, Mahajan A, Fujimura O, Boyle NG, Shivkumar K. Radiofrequency current delivery via transseptal needle to facilitate septal puncture. Heart Rhythm. 2007 Dec;4(12):1573-6. doi: 10.1016/j.hrthm.2007.07.008. Epub 2007 Jul 14. No abstract available. PMID 17997362
- [Background] Justino H, Benson LN, Nykanen DG. Transcatheter creation of an atrial septal defect using radiofrequency perforation. Catheter Cardiovasc Interv. 2001 Sep;54(1):83-7. doi: 10.1002/ccd.1244. PMID 11553955
- [Background] Smelley MP, Shah DP, Weisberg I, Kim SS, Lin AC, Beshai JF, Burke MC, Knight BP. Initial experience using a radiofrequency powered transseptal needle. J Cardiovasc Electrophysiol. 2010 Apr;21(4):423-7. doi: 10.1111/j.1540-8167.2009.01656.x. Epub 2009 Nov 17. PMID 19925604
- [Background] Sakata Y, Feldman T. Transcatheter creation of atrial septal perforation using a radiofrequency transseptal system: novel approach as an alternative to transseptal needle puncture. Catheter Cardiovasc Interv. 2005 Mar;64(3):327-32. doi: 10.1002/ccd.20284. PMID 15736263
- [Background] Crystal MA, Mirza MA, Benson LN. A radiofrequency transseptal needle: initial animal studies. Catheter Cardiovasc Interv. 2010 Nov 1;76(5):769-73. doi: 10.1002/ccd.22600. PMID 20506170
- [Derived] Hsu JC, Badhwar N, Gerstenfeld EP, Lee RJ, Mandyam MC, Dewland TA, Imburgia KE, Hoffmayer KS, Vedantham V, Lee BK, Tseng ZH, Scheinman MM, Olgin JE, Marcus GM. Randomized trial of conventional transseptal needle versus radiofrequency energy needle puncture for left atrial access (the TRAVERSE-LA study). J Am Heart Assoc. 2013 Sep 17;2(5):e000428. doi: 10.1161/JAHA.113.000428. PMID 24045120

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January 2011 and November 2012, 72 patients were randomized to 1 of 2 transseptal needle groups.
Pre-assignment Details: 139 patients were assessed for eligibility; 61 declined to participate, 3 met exclusion criteria, 3 did not enroll for other reasons.
Groups:
- Radiofrequency Energy Needle: Transseptal access using a radiofrequency energy needle. Participants for whom puncture failed crossed over to the other intervention; all study analyses were performed on an intention-to-treat basis.
- Mechanical Needle: Transseptal access using a mechanical (Brockenbrough) needle. Participants for whom puncture failed crossed over to the other intervention; all study analyses were performed on an intention-to-treat basis.
Period: Overall Study
Arm/Group | Radiofrequency Energy Needle | Mechanical Needle
Started | 36 | 36
Completed | 36 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: per protocol
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiofrequency Energy Needle | Mechanical Needle | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (11.3) | 61.1 (11.7) | 60.5 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 25 | 23 | 48
Region of Enrollment [Number; unit: participants]
  United States | 36 | 36 | 72
Previous stroke or transient ischemic attack (TIA) [Number; unit: participants]
  Previous stroke or TIA | 2 | 3 | 5
  No previous stroke or TIA | 34 | 33 | 67
Indication for transseptal puncture [Number; unit: participants]
  Atrial fibrillation | 35 | 35 | 70
  Accessory pathway | 1 | 1 | 2
History of transseptal puncture [Number; unit: participants]
  Previous transseptal puncture | 12 | 10 | 22
  No previous transseptal puncture | 24 | 26 | 50

OUTCOME MEASURES:

1. Primary Outcome: Transseptal Access Procedure Time
Description: Total amount of procedure time, from the beginning of the transseptal procedure until left atrium (LA) access is obtained in each patient. Participants for whom puncture failed crossed over to the other Intervention. Analysis performed on an intention-to-treat basis.
Time Frame: Day of procedure
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Radiofrequency Energy Needle | Mechanical Needle
Number analyzed (Participants) | 36 | 36
minutes | 2.3 [1.7 to 3.8] | 7.3 [2.7 to 14.1]
Statistical Analysis 1: Comparison: Radiofrequency Energy Needle vs Mechanical Needle; Sample size of 72 was targeted to achieve 80% power to detect a 5-minute reduction in transseptal access procedure time (assuming a standard deviation of 7.5 minutes), using a 2-sided alpha of 0.05, with the primary analysis done on an intention-to-treat basis; Test type: Superiority or Other; p = 0.005, t-test, 2 sided — Statistical tests were 2-sided and considered significant if they yielded a p<0.05

2. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety
Time Frame: During or immediately after procedure, up to 1 day after procedure. On average, up to 1 day after the procedure.
Measure: Number; unit: participants
Arm/Group | Radiofrequency Energy Needle | Mechanical Needle
Number analyzed (Participants) | 36 | 36
participants | 1 | 1

3. Secondary Outcome: Performance of the Assigned Needle Type
Description: Failure to achieve transseptal access with the assigned needle type resulted in crossover because of an inability to puncture the interatrial septem despite forward pressure and tenting, leading to concern that further effort might lead to perforation of the free (lateral) LA wall.
Time Frame: at time of procedure
Measure: Number; unit: participants
Groups:
- Radiofrequency Energy Needle: Transseptal access using a radiofrequency energy needle
- Mechanical Needle: Transseptal access using a mechanical (Brockenbrough) needle
Arm/Group | Radiofrequency Energy Needle | Mechanical Needle
Number analyzed (Participants) | 36 | 36
participants
  Success of assigned needle type | 36 | 26
  Failure of assigned needle type | 0 | 10
Statistical Analysis 1: Comparison: Radiofrequency Energy Needle vs Mechanical Needle; Test type: Superiority or Other; p < 0.001, Chi-squared — Statistical tests were 2-sided and considered significant if they yielded a p<0.05

4. Secondary Outcome: Plastic Dilator Shavings
Description: In ex vivo pre-procedural testing, the assigned transseptal needle was advanced through the plastic dilator and sheath, and the presence of grossly visible plastic shavings after introduction of the needle through the dilator and long sheath was recorded.
Time Frame: immediately prior to procedure
Population: The assigned needle for each participant was analyzed prior to the procedure
Measure: Number; unit: Needles
Units Other Than Participants: Assigned needles
Arm/Group | Radiofrequency Energy Needle | Mechanical Needle
Number analyzed (Participants) | 36 | 36
Number analyzed (Assigned needles) | 36 | 36
Needles | 0 | 12
Statistical Analysis 1: Comparison: Radiofrequency Energy Needle vs Mechanical Needle; Test type: Superiority or Other; p < 0.001, Chi-squared — Statistical tests were 2-sided and considered significant if they yielded a p<0.05

ADVERSE EVENTS:
Time Frame: During or immediately after procedure, up to 1 day after procedure. On average, up to 1 day after the procedure.
Description: All patients were monitored for both intraprocedural complications and postprocedural complications until discharge. Participants for whom puncture failed crossed over to the other intervention; all study analyses were performed on an intention-to-treat basis.
Groups:
- Radiofrequency Energy Needle (RF): Transseptal access using a radiofrequency energy needle. Participants for whom puncture failed crossed over to the other intervention; all study analyses were performed on an intention-to-treat basis.
Arm/Group | Radiofrequency Energy Needle (RF) | Mechanical Needle
Serious Adverse Events (participants affected / at risk) | 1/36 | 1/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiofrequency Energy Needle (RF) (N=36) | Mechanical Needle (N=36)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) — Pericardial effusion detected by intracardiac echocardiography (ICE) after conclusion of the LA ablation procedure, 3 hours after the transseptal puncture.
Transient ischemic attack (Vascular disorders) | 0 (0) | 1 (1) — transient ischemic attack with brain magnetic resonance imaging consistent with embolic etiology

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes